CLINICAL TRIAL: NCT02608372
Title: Effect of Brown Seaweeds on Glycaemia, Gastric Emptying, and Appetite: A Randomized, Controlled Crossover Meal Study
Brief Title: Brown Seaweeds Effect on Glucose Tolerance and Appetite Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Ministry of Education, Malaysia (Other Government); Universiti Malaysia Pahang (Other)
Responsible Party: Principal Investigator, Professor Lars Ove Dragsted, Professor, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: M221
Record Dates: First submitted 2015-11-14; First posted 2015-11-18 (Estimated); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: High Blood Glucose
Keywords: Seaweed; Insulin; Glucose tolerance; C-peptide; Appetide; Metabolomics
MeSH Terms: conditions — Hyperglycemia; Insulin Resistance

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Sequence A (Experimental): The meal study was performed with Laminaria digitata (LD), Undaria pinnatifida (UP) or pea protein drink (CTR) in the sequence LD-UP-CTR
  Interventions: Other: LD; Other: UP; Other: CTR
- Sequence B (Experimental): The meal study was performed with Laminaria digitata (LD), Undaria pinnatifida (UP) or pea protein drink (CTR) in the sequence LD-CTR-UP
  Interventions: Other: LD; Other: UP; Other: CTR
- Sequence C (Experimental): The meal study was performed with Laminaria digitata (LD), Undaria pinnatifida (UP) or pea protein drink (CTR) in the sequence UP-LD-CTR
  Interventions: Other: LD; Other: UP; Other: CTR
- Sequence D (Experimental): The meal study was performed with Laminaria digitata (LD), Undaria pinnatifida (UP) or pea protein drink (CTR) in the sequence UP-CTR-LD
  Interventions: Other: LD; Other: UP; Other: CTR
- Sequence E (Experimental): The meal study was performed with Laminaria digitata (LD), Undaria pinnatifida (UP) or pea protein drink (CTR) in the sequence CTR-LD-UP
  Interventions: Other: LD; Other: UP; Other: CTR
- Sequence F (Experimental): The meal study was performed with Laminaria digitata (LD), Undaria pinnatifida (UP) or pea protein drink (CTR) in the sequence CTR-UP-LD
  Interventions: Other: LD; Other: UP; Other: CTR

INTERVENTIONS:
Other: LD — Participants ingested 5 g of Laminaria digitata followed by 30 g of corn starch mixed with 200 mL of water.
Other: UP — Participants ingested 5 g of Undaria pinnatifida followed by 30 g of corn starch mixed with 200 mL of water.
Other: CTR — Participants ingested 30 g of corn starch and 1 g of pea protein powder mixed with 200 mL of water.

SUMMARY:
The project is a randomized, 3-way, blinded crossover trial in which 20 healthy, fasted participants consume meals with 30 g of a linear corn starch and 5 g of one of the seaweeds, Laminara digitata or Undaria pinnatifida or a pea protein control. The primary aim is to investigate whether the brown seaweeds affect the postprandial glucose Area Under the Curve (AUC). Stomach emptying, insulin, C-peptide, appetite-regulating hormones (oxyntomodulin, glucagon, GLP-1 and PYY), and specific metabolites from the seaweeds in the urine and plasma as well as subjective satiety are also analyzed.

DETAILED DESCRIPTION:
Brown seaweeds may contain bioactive compounds as they contain secondary plant metabolites, including flavonoids and other phenolic compounds as well as carotenoids. Dietary fibre is the major component of brown seaweeds, mainly composed from laminarans, alginates, fucans and cellulose. Several dietary fibers and secondary plant metabolites have been shown to have an impact on health and more specifically on glycemic control. Therefore, the aim of this study was to investigate whether two selected brown seaweeds have an effect on the postprandial glucose response to a starch load as well as several secondary measures, including appetite responses.

In a controlled crossover trial, 20 healthy fasted participants consumed 5 g of either Laminaria digitata (LD) or Undaria pinnatifida (UP) or 1 g of pea protein (CTR). The volunteers concomitantly ingested 200 mL of a drink with corn starch. Blood samples were drawn at baseline, as well as 20, 40, 60, 90, 120 and 180 min after the meal. Differences in glucose, insulin, C-peptide, plasma incretin concentrations, and insulin sensitivity index (ISI) were analyzed and appetite was scored by a visual analogue scale and a subsequent ad libitum test meal.

ELIGIBILITY:
Inclusion Criteria:

BMI 20-25 kg/m2. Waist circumference < 102 cm. Non-smoking. Like (can tolerate) seaweed, pasta, meat sauce as these foods are part of the test meal.

Can tolerate paracetamol (Pinex, Actavis, Denmark).

Exclusion Criteria:

Systemic infections, psychiatric or metabolic diseases, and any clinical condition, chronic or frequent use of medication (including blood thinners, excluding contraceptives), smoking (throughout the trial and 12 months before the start of the experiment), blood donations during or in the month leading up to the study period, elite athletes (> 10 hours of hard exercise / week, self-reported), high intake of alcohol (defined as a weekly intake of > 7 units for women and > 14 units for men), have or have had a drug addiction, participation in other scientific studies during the study period, lactating, pregnancy or ongoing planning of pregnancy, and vegetarianism or veganism.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-05; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Plasma glucose Area Under the Curve (Glucose AUC) | 0- 180 min
  The area under the plasma glucose concentration curve was calculated from 0-180 min after 30 g of corn starch was ingested.

SECONDARY OUTCOMES:
Plasma glucose concentrations | 20, 40, 60, 90, 120 and 180 min
  Changes in the glucose concentrations determined by a mixed model analysis and subsequently at each time point with time 0 as a co-variate.
Serum Insulin Area Under the Curve | 0-180 min
  Area Under the Curve (AUC) for serum insulin.
Serum Insulin concentrations | : 20, 40, 60, 90, 120 and 180 min
  Changes in the insulin concentrations determined by a mixed model analysis and subsequently at each time point with time 0 as a co-variate.
ISI (0-180) | 0-180 min
  Matsuda's Insulin Sensitivity Index
Serum C-peptide Area Under the Curve | 0-180 min
  Area Under the Curve (AUC) for serum C-peptide.
Serum C-peptide concentrations | 20, 40, 60, 90, 120 and 180 min
  Changes in the C-peptide concentrations determined by a mixed model analysis and subsequently at each time point with time 0 as a co-variate.
Plasma GLP-1 Area Under the Curve | 0-180 min
  Area Under the Curve (AUC) for plasma GLP-1.
Plasma GLP-1 concentrations | 20, 40, 60, 90, 120 and 180 min
  Changes in the plasma GLP-1 concentrations determined by a mixed model analysis and subsequently at each time point with time 0 as a co-variate
Subjective appetite scores assessed by visual analogue scale (VAS) | 0-180 min
  Area Under the Curve (AUC) for all VAS outcomes (satiety, hunger, fullness, prospective food consumption and comfort)
Subjective appetite scores assessed by visual analogue scale (VAS) | 20, 40, 50, 70, 100, 130 and 180 min
  Changes in VAS outcomes (satiety, hunger, fullness, prospective food consumption and comfort), determined by a mixed model analysis and subsequently at each time point with time 0 as a co-variate

OTHER OUTCOMES:
Metabolic profile in urine | 0-24 hrs
  Untargeted metabolic profile of urine samples measured in all samples collected before the meal and postprandially from 0-90 min, 90-180 min as well as in samples collected up to 24 hours later. The totality of the profiles is used to explore for changes after baseline as detected by multivariate statistics (PLS-DA) after dividing the data into a training and test set. Contrasts between each of the treatment groups and the placebo group will be assessed using the receiver-operator characteristics (ROC curves) comparing the training and test set.
Metabolic profile in plasma | 0-180 min
  Untargeted metabolic profile of plasma measured in all samples collected before the meal and postprandially from 0-180 min. The totality of the profile is used to explore for changes after baseline as detected by multivariate statistics (PLS-DA) after dividing the data into a training and test set. Contrasts between each of the treatment groups and the placebo group will be assessed using the receiver-operator characteristics (ROC curves) comparing the training and test set.

CONTACTS AND LOCATIONS:
Overall Officials: Lars O Dragsted, PhD, Principal Investigator — University of Copenhagen
Locations (1):
- Department of Nutrition, Exercise and Sports, University of Copenhagen, Frederiksberg, Denmark

REFERENCES:
- [Derived] Zaharudin N, Tullin M, Pekmez CT, Sloth JJ, Rasmussen RR, Dragsted LO. Effects of brown seaweeds on postprandial glucose, insulin and appetite in humans - A randomized, 3-way, blinded, cross-over meal study. Clin Nutr. 2021 Mar;40(3):830-838. doi: 10.1016/j.clnu.2020.08.027. Epub 2020 Aug 31. PMID 32917417